CLINICAL TRIAL: NCT03818425
Title: Motivation and Barriers for Exercise in Patients With Anxiety or Posttraumatic Stress Disorder
Status: Completed | Type: Observational
Sponsor: Universitaet Innsbruck (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 256913
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Exercise; Motivation
Keywords: Anxiety; Posttraumatic Stress Disorder
MeSH Terms: conditions — Motor Activity; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical Population: In- and Out-Patients diagnosed with depression (F32, F33), anxiety disorder (F40, F41; ICD-10) or posttraumatic stress disorder (F43.1; ICD-10)
- Healthy Controls: Subjects with no previous or actual mental disorder

SUMMARY:
Relevance and Aim: There has been increasing research interest in sport preferences and motivational factors as well as barriers that restrain from engaging in sport activities in people suffering from mental illnesses. Anxiety disorders are one of the leading mental disorders worldwide. Exercise has previously shown anxiolytic effects and is discussed as an adjunctive treatment option in clinical practice. This study aims to depict motivation and barriers in patients with anxiety or posttraumatic stress disorders.

Design and Participants: Observational study of patients diagnosed with anxiety disorder or posttraumatic stress disorder (ICD-10)

Measurements: Structured questionnaire compounded of validated scales for current physical activity, sport motivation, exercise preferences, perceived barriers , self-efficacy, social support for physical activity, motivation,enjoyment, quality of life as well as sociodemographic data.

Duration: The questionnaire will require approximately 20 minutes, the overall duration is 3 months. Personal assistance for completing the questionnaire will be provided if necessary.

ELIGIBILITY:
Inclusion Criteria:

* In- and out-patients with a diagnosed anxiety or posttraumatic stress disorder (F40, F41, F43.1; ICD-10)
* 18 to 65 years

Exclusion Criteria:

* acute psychosis or suicidal behaviour
* cognitive deficits
* problems with German language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of outpatient department and inpatients of the Medical Hospital Innsbruck, Department of Psychiatry and Psychosomatic will be selected by clinical professionals according to inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Physical activity | 5 minutes
  self reported, actual physical activity, measured by the International Physical Activity Questionnaire Short Form, IPAQ-SF; Craig et al., 2003
Sport motivation | 5 minutes
  measured by the Exercise Motivation Inventory, EMI-2; Markland & Hardy,1993
Perceived barriers | 5 minutes
  measured by 12 questions referring to Ussher, Stanbury, Cheeseman & Faulkner, 2007
Self-efficacy for physical activity | 1 minute
  single item question according to Ussher, Stanbury, Cheeseman & Faulkner, 2007
Social support for physical activity | 1 minute
  single item question according to Ussher, Stanbury, Cheeseman & Faulkner, 2007
Motivation for physical activity | 1 minute
  single item question according to Ussher, Stanbury, Cheeseman & Faulkner, 2007
Enjoyment of physical activity | 1 minute
  single item question according to Ussher, Stanbury, Cheeseman & Faulkner, 2007

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kopp, PhD, Prof., Study Chair — Department of Sport Science, University of Innsbruck; Barbara Sperner-Unterweger, MD, Prof., Study Director — Department of Psychosomatics, Medical University of Innsbruck
Locations (1):
- University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bichler CS, Niedermeier M, Gufler A, Galffy M, Sperner-Unterweger B, Kopp M. A case-control study on physical activity preferences, motives, and barriers in patients with psychiatric conditions. Compr Psychiatry. 2021 Nov;111:152276. doi: 10.1016/j.comppsych.2021.152276. Epub 2021 Sep 23. PMID 34600310